CLINICAL TRIAL: NCT07364838
Title: A Phase 1 Clinical Trial to Evaluate the Effect of Food on the Safety, Pharmacokinetics and Pharmacodynamics Characteristics of DW4421 in Healthy Adult Volunteers
Brief Title: Study to Evaluate the Effect of Food on the Pharmacokinetics and Pharmacodynamics Characteristics in Healthy Adult Volunteers
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Daewon Pharmaceutical Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: DW4421-101
Record Dates: First submitted 2025-12-22; First posted 2026-01-23 (Actual); Last update posted 2026-01-23 (Actual); Status verified 2025-12

CONDITIONS: GERD (Gastroesophageal Reflux Disease)
MeSH Terms: conditions — Gastroesophageal Reflux

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Sequence A (Experimental): Cross-over
  Interventions: Drug: DW4421
- Sequence B (Experimental): Cross-over
  Interventions: Drug: DW4421

INTERVENTIONS:
Drug: DW4421 — DW4421 on fasted or fed condition

SUMMARY:
A Randomized, Open-label, Oral in healthy volunteers

ELIGIBILITY:
Inclusion Criteria:

* Healthy Volunteers who are ≥19 years old
* Body weight ≥50.0 kg and BMI between 18.0 and 30.0 kg/m2

Exclusion Criteria:

* Clinically significant Medical History
* In the case of women, pregnant(Urine-HCG positive) or lactating women

Ages: 19 Years to 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 24 (Actual)
Dates: Start 2024-11-21 (Actual); Primary Completion 2025-04-08 (Actual); Study Completion 2025-04-08 (Actual)

PRIMARY OUTCOMES:
Peak Plasma Concentration (Cmax) | up to 48 hours
  Cmax of DW4421
Area under the plasma concentration versus time curve (AUC) | up to 48 hours
  AUC of DW4421

CONTACTS AND LOCATIONS:
Locations (1):
- Chungbuk National University Hospital, Cheongju-si, South Korea